CLINICAL TRIAL: NCT04579003
Title: Effect of Shoulder Mobilization and Mobilization With Movement on Sub Acromial Space in Shoulder Impingement.
Brief Title: Mobilization and Mobilization With Movement Effect on Sub Acromial Space in Impingement Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00692 Aneela Ghafoor
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Impingement Syndrome
Keywords: Impingement syndrome; Mobilization; Mobilization with movement; Sub acromial space
MeSH Terms: interventions — Movement

STUDY DESIGN:
Intervention Model Description: Both groups were treated simultaneously with their specified treatment techniques within given duration.
Who Masked: Participant
Masking Description: Participants did not know which treatment techniques are given in the specified groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization (Experimental): Mobilization, heat application, ultrasound, TENS
  Interventions: Other: Mobilization
- Mobilization with movement (Active Comparator): Mobilization with movement, heat application, ultrasound, TENS
  Interventions: Other: Mobilization with movement

INTERVENTIONS:
Other: Mobilization — Moist hot pack for 10 mins/1 set/ 6 consecutive days, Ultrasound for 5 mins/1 set/ 6 consecutive days, TENS on shoulder region for 10 mins/1 set/ 6 consecutive days, Shoulder mobilization posterolateral glide for 30 secs with 30 secs rest for 5 mins.
  A total of 6 consecutive sessions were given each consisting of 30 mins.
  Arms: Mobilization
Other: Mobilization with movement — Moist hot pack for 10 mins/1 set/ 6 consecutive days, Ultrasound for 5 mins/1 set/ 6 consecutive days, TENS on shoulder region for 10 mins/1 set/ 6 consecutive days, Shoulder mobilization with movement (MWM) 10 repetitions with 30 secs rest for 5 mins.
  A total of 6 consecutive sessions were given each consisting of 30 mins.
  Arms: Mobilization with movement

SUMMARY:
Mobilization and mobilization with movement both treatment techniques are effective in impingement syndrome.The objective of our study is to compare the effects of shoulder mobilization and mobilization with movement on subacromial space in impingement syndrome.

DETAILED DESCRIPTION:
A study was conducted in 2016 to determine the effect of MWM in Impingement syndrome on sub acromial space, pain and disability. In this study,15 patients diagnosed with sub acromial impingement were selected and treated for six sessions. MWM posterolateral glide was the intervention selected. The results showed the p value of <0.00001 for pre and post treatment sessions of MWM in patients with Impingement syndrome. According to the results it was concluded that in terms of decreasing the pain and disability as well as increasing the acromiohumeral distance MWM is effective treatment for impingement syndrome.

An RCT was conducted in 2016 to find out the effect of posterolateral glide MWM on pain, strength of shoulder muscles and upward rotation of scapula. 31 patients were allocated to a group performing exercises actively and other group who received posterolateral glides MWM. The results suggested that MWM was effective intervention in decreasing pain on VAS and improving strength of external rotators.

A study was conducted in 2013 to compare the effects of supervised exercise with and without manual therapy for impingement syndrome.The results showed marked differences in reducing pain and increasing ROM and strength of rotator muscles in group that received supervised exercise with manual therapy. So it was concluded that manual therapy with exercise program is effective in decreasing pain and improving ROM than exercises alone in impingement syndrome.

A study was conducted to compare the effects of mobilization with movement and mobilization with therapeutic exercises in patients of subacromial impingement. The results are suggestive that shoulder mobilization and MWM with exercises result in more reduction of pain and improved AROM.

A RCT was conducted to compare the effectiveness of joint and soft tissue mobilization techniques and self-training program. The results of this study showed that patient who received manual therapy showed significant differences. So it was concluded that joint mobilization is effective intervention for patients with impingement syndrome.

Studies have been conducted in the past on effect of mobilization and mobilization with movement on shoulder impingement but they did not report their effect on sub acromial space in impingement syndrome using musculoskeletal ultrasound and the comparison of both techniques.

The purpose of this study is to find out the effects of mobilization and mobilization with movement on sub acromial space using musculoskeletal ultrasound in impingement syndrome and compare their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Impingement Syndrome Screening using Neer Impingement Test, Hawkin Kennedy Test.
* Patients with impingement syndrome in acute phase.

Exclusion Criteria:

* Frozen Shoulder
* Thoracic Outlet Syndrome
* Cervical Radiculopathy
* Any Fracture or dislocation of shoulder girdle.
* Diabetic Patients.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
Sub acromial Space | 6th day
  Changes from baseline, for measuring sub acromial space, patients were seated with arm resting at the side with fully extended elbow, trunk in neutral position and ultrasound images were taken using linear transducer probe. The ultrasound transducer was positioned on the shoulder over the acromion and humeral head. AHD was measured using onscreen calipers by finding superior aspect of head of humerus and inferior aspect of acromion (between apex of greater tubercle of humerus and inferior edge of acromial process). Three readings were taken which then averaged for a single reading.

SECONDARY OUTCOMES:
Supraspinatus Tendon Thickness | 6th day
  Changes from baseline, Transducer was placed on shoulder over subacromial space with the notch diagonally facing down towards the belly button, measured in transverse view lateral to the biceps tendon of long head.
Numeric Pain Rating Scale | 6th day
  Changes from baseline, Numeric pain rating scale is a scale from 0 to 10. 0 indicating no pain and 10 indicating worse pain.
Range of motion ( ROM) | 6th day
  Changes from baseline, shoulder ROM were taken using goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, Phd, Principal Investigator — Riphah International University
Locations (1):
- Max Rehab & Physical Therapy Centre G-8 Markaz, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ajit D, Shika S. Effects of Mobilization with Movement (MWM) in Shoulder Impingement Syndrome Patients on Acromiohumeral Distance using Ultrasonography. Journal of Exercise Science & Physiotherapy. 2016;12(2).
- [Background] Neelapala YR, Reddy YRS, Danait R. Effect of mulligan's posterolateral glide on shoulder rotator strength, scapular upward rotation in shoulder pain subjects-a randomized controlled trial. Journal of Musculoskeletal Research. 2016;19(03):1650014.
- [Background] Bang MD, Deyle GD. Comparison of supervised exercise with and without manual physical therapy for patients with shoulder impingement syndrome. J Orthop Sports Phys Ther. 2000 Mar;30(3):126-37. doi: 10.2519/jospt.2000.30.3.126. PMID 10721508
- [Background] Kachingwe AF, Phillips B, Sletten E, Plunkett SW. Comparison of manual therapy techniques with therapeutic exercise in the treatment of shoulder impingement: a randomized controlled pilot clinical trial. J Man Manip Ther. 2008;16(4):238-47. doi: 10.1179/106698108790818314. PMID 19771196